CLINICAL TRIAL: NCT03869944
Title: Elimination of Paediatric HIV-1 Infection: Evaluation of the Prevention Programme and Rescue Intervention Based on the Expanded Programme on Immunization (EPI). ANRS 12388 PREVENIR-PEV Study.
Brief Title: Preventing Childhood HIV: Rescue Intervention. ANRS 12388 PREVENIR-PEV
Acronym: PREVENIR-PEV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre Muraz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 12388 PREVENIR-PEV
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: HIV-1
Keywords: HIV-1; PMTCT; Point of Care; PrEP; Burkina Faso; Expanded Program of Immunization (EPI)
MeSH Terms: interventions — Lamivudine

STUDY DESIGN:
Intervention Model Description: Phase II trial, non-randomized, open-label, mono-country and multi-center trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Lamivudine Oral Solution
  Interventions: Drug: Lamivudine Oral Solution

INTERVENTIONS:
Drug: Lamivudine Oral Solution — During the EPI-2 visit, HIV-1 negative children of mothers with a unsuppressed plasma HIV-1 VL (≥ 1000 copies/mL) will be initiated on PrEP, lamivudine syrup (7.5 mg twice daily if 2 to 4 kg; 25 mg twice a day if weight <8 kg; and 50 mg twice a day if weight >8 kg) for 10 months, until the child is 12 months old. A monitoring on the mother's VL and child's diagnosis will take place at 6 and 12 months.
  Mothers with unsuppressed plasma HIV-1 VL (< 1000 copies/mL) and HIV-1 negative children will not be offered PrEP but the mother's VL and child diagnosis will be monitored at 6 and 12 months: If the VL is ≥ 1000 copies/mL, the child will be initiated on PrEP until the child is 12 months old.
  Children infected with HIV-1 will be referred to the National Program for immediate ART.

SUMMARY:
The second visit of the Expanded Programme of Immunization when the child is 2 months old (EPI-2) represents a unique opportunity to link the EPI and PMTCT programmes and to introduce preventive and therapeutic rescue interventions in order to 1) Assess the efficacy of the PMTCT cascade up to 2 months postpartum; 2) Allow at least 80% of HIV-1-infected infants identified at the second EPI visit who were not involved in HIV care to initiate ARVs at the earliest, but no later than 2 months after confirmation of HIV diagnosis; 3) Reduce HIV-1 transmission to less than 3% between 2 and 12 months among exposed children who completed the second EPI visit

DETAILED DESCRIPTION:
The WHO recommendation of lifelong antiretroviral therapy (ART) for all HIV-infected pregnant or breastfeeding women represents a major advance for universal access to HIV care but this strategy alone may not be sufficient to eliminate pediatric HIV in the communities.

Presently, the impact of prevention of mother-to-child HIV transmission (PMTCT) programs in the communities is unclear. There is also no available rescue intervention able to identify postpartum women at high risk of transmission in order to offer them adequate HIV care and prevent HIV acquisition by their breastfed infants.

We hypothesize that the second visit for routine vaccination (Expanded Program of Immunization visit 2, EPI-2) represents a unique opportunity to link EPI and PMTCT programs and introduce rescue preventive and therapeutic interventions.

The study will assess the efficacy of the PMTCT cascade up to 2 months post-partum for all mothers attending the EPI-2 (Component 1). For Component 1, the target population will be all 32,100 women participating in EPI-2 and verbally consenting to participate to evaluate the PMTCT program up to 2 months postpartum.

The consent form for component 2 will be proposed to all HIV positive mothers of component 1 who meet the inclusion and non-inclusion criteria. HIV-1 viral load measurement of the mothers and the detection of HIV-1 DNA in their children will be assessed. Children infected with HIV-1 will be referred for immediate ART initiation.

For Component 2 - phase IIb trial (N = 300 mother-infant pairs) - the target population will be HIV positive breastfeeding mothers aged 15 years or older with a child whose tests so far do not reveal the existence of infection (at EPI-2 visit) to assess the effectiveness of a rescue intervention for Prevention of Mother-to-Child Transmission of HIV up to 12 months of age.

The target population to receive PrEP (lamivudine) until 12 months of age (or until confirmed end of breastfeeding) will be women with unsuppressed HIV-1 infection (≥1000 copies of HIV-1 RNA/ml) with a child whose tests to date (EPI-2 visit) do not reveal the existence of infection.

HIV-1 infected women with suppressed (<1000 copies of HIV-1 RNA/ml) viral load at the time of the EPI-2 visit will be followed at 6 and 12 months. If at 6 months the mother become virally unsuppressed, her child will receive ARV medication up to 12 months of age (or the confirmed end of breastfeeding) to prevent infection.

The control group does not apply to this study. The overall mother-to-child transmission rate is the WHO target for the elimination of paediatric HIV-1: 5% at one year of life (consistent with a 3% postnatal transmission rate between 2 and 12 months of age of the child).

ELIGIBILITY:
For HIV+ women who give consent, the measurement of their HIV-1 viral load and the detection of HIV-1 DNA in their children will be assessed.

Inclusion Criteria:

A mother-child couple will be included in the Phase IIb trial if the child:

* is a singleton
* is breastfed at about 2 months and the mother intends to continue breastfeeding for at least 4 months (until her child is 6 months old)
* has a POC HIV-1 PCR negative test at about 2 months of age
* has a mother who:
* accompanies him to visit 2 of the EPI
* is over 20 years of age or over or is a minor from the age of 15 and is accompanied by a referent adult of his/her choice representing his/her interests (parent, family member or guardian, member of an association, etc.)
* has been confirmed to be infected with HIV-1 (with or without HIV-2)
* signature of the consent to participate
* for the mother signed by herself and a witness (if illiterate) and/or a referent adult (if under 20 years of age)
* for the child: consent must be signed by both parents unless the mother exercises parental authority alone or if obtaining the father's consent is likely to endanger the mother and her child.

Exclusion Criteria:

A mother-child couple will not be included in the Phase IIb trial if the child:

* exhibits DAIDS grade 3 or 4 clinical symptoms or biological anomalies for adverse events on the day of inclusion
* has a severe congenital malformation
* has a known allergy to the study drug or its components
* is taking emtricitabine concomitantly
* has a mother:
* living outside the study area or planning to move from the area within the next 12 months
* participating in another clinical trial on the day of inclusion

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — HIV-1-positive breastfeeding mothers of HIV-1-negative children (female or male)
Enrollment: 97 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Prevention of HIV-1 transmission from HIV-1-positive mothers to their breastfeeding children | 12 months
  Postnatal HIV-1 transmission rates at 12 months in infants exposed to HIV-1 through breastfeeding.

SECONDARY OUTCOMES:
Efficacy of PMTCT cascade - mother | 2 months
  Proportion of EPI-2 women who did not attend PMTCT clinic at least once during pregnancy (as per the records in the antenatal care clinics): Proportion who received an HIV-1 test in the three previous months (as per the records in the antenatal care clinics); Proportion of women infected with HIV-1 and Proportion with undetectable plasma viral load (<1000 copies of HIV RNA/mL) (as per the results obtained with the Point of Care HIV-1 PCR Viral Load in the study), Proportion of mothers who started antiretroviral treatment during pregnancy or after delivery (as per the records in the antenatal care clinics)
Efficacy of PMTCT cascade - child | 2 months
  Proportion of babies with HIV-1 PCR positive (as per the results obtained with the Point of Care HIV-1 PCR Qualitative in the study); Proportion of HIV-1-infected babies engaged in HIV care at 2 months (i.e. initiated on antiretroviral treatment) (as per the data collected at the study sites following diagnosis by Point of Care HIV-1 PCR).
Access to ART for HIV-1-positive children | 6 months
  Proportion of HIV-infected infants identified at the second EPI visit who were not engaged in HIV care at that time, who will be placed on ART within two months of that visit, or if they are infected during follow-up within two months of diagnosis.
Number of Adverse Events Grade 3 and 4 in the prevention of HIV-1 via breastfeeding [Safety of lamivudine] | 12 months
  • Adverse event rates at 12 months, including deaths and Grade 3 or 4 events on the pediatric DAIDS scale in uninfected children exposed to HIV

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Van de Perre, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Paulin Fao, Bobo-Dioulasso, Burkina Faso

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nagot N, Kankasa C, Tumwine JK, Meda N, Hofmeyr GJ, Vallo R, Mwiya M, Kwagala M, Traore H, Sunday A, Singata M, Siuluta C, Some E, Rutagwera D, Neboua D, Ndeezi G, Jackson D, Marechal V, Neveu D, Engebretsen IMS, Lombard C, Blanche S, Sommerfelt H, Rekacewicz C, Tylleskar T, Van de Perre P; ANRS 12174 Trial Group. Extended pre-exposure prophylaxis with lopinavir-ritonavir versus lamivudine to prevent HIV-1 transmission through breastfeeding up to 50 weeks in infants in Africa (ANRS 12174): a randomised controlled trial. Lancet. 2016 Feb 6;387(10018):566-573. doi: 10.1016/S0140-6736(15)00984-8. Epub 2015 Nov 19. PMID 26603917
- [Derived] Mennecier A, Sakana BLD, D'Ottavi M, Tassembedo S, Moles JP, Kania D, Taofiki AO, Kadeba FE, Diallo I, Eymard-Duvernay S, Meda N, Mosqueira B, Fao P, Nagot N; PREVENIR-PEV Study Group; Vande Perre P. An optimized strategy triggered at the 2nd immunization visit to prevent HIV acquisition by breastfeeding: a phase 2 trial in Burkina Faso (PREVENIR-PEV). BMC Infect Dis. 2024 Sep 20;24(1):1014. doi: 10.1186/s12879-024-09910-z. PMID 39300364
- [Derived] Mennecier A, Kankasa C, Fao P, Moles JP, Eymard-Duvernay S, Mwiya M, Kania D, Chunda-Liyoka C, Sakana L, Rutagwera D, Tassembedo S, Wilfred-Tonga MM, Mosqueira B, Tylleskar T, Nagot N, Van de Perre P; ANRS 12397 Study group. Design and challenges of a large HIV prevention clinical study on mother-to-child transmission: ANRS 12397 PROMISE-EPI study in Zambia and Burkina Faso. Contemp Clin Trials. 2021 Jun;105:106402. doi: 10.1016/j.cct.2021.106402. Epub 2021 Apr 17. PMID 33872801